CLINICAL TRIAL: NCT03958578
Title: The Effect of Preoperative Anxiety on Duration and Efficacy of Motor and Sensory Block in Spinal Anesthesia
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Yadigar Yılmaz, Medical Doctor, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Other Study IDs: OKMEYDANI EAH 48670771-514.10
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Spinal anaesthesia results in blockade of sympathetic efferent neurones. Patients with higher baseline sympathetic activation have been shown to have more marked hypotension after spinal anaesthesia. Anxiety causes generalized sympathetic activation. It was aimed to find the effect of preoperative anxiety on the duration and efficacy of neuraxial anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 55 years.
* ASA I-II
* BMI 18-25

Exclusion Criteria:

* Major surgery

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: It is planned to enroll healthy individuals undergoing elective surgery under spinal anaesthesia.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory questionnaire | 20-30 minutes.
  State-Trait Anxiety Inventory questionnaire is a direct psychological assessment of preoperative anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Yadigar Yılmaz, Istanbul, Turkey (Türkiye)